CLINICAL TRIAL: NCT02706483
Title: An Open Label, Long Term Safety and Tolerability Study of Plecanatide in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Long Term Safety Study of Plecanatide
Acronym: IBS-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP304203-06
Record Dates: First submitted 2016-02-29; First posted 2016-03-11 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — plecanatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plecanatide (Experimental): Plecanatide 6.0 mg tablets
  Interventions: Drug: Plecanatide

INTERVENTIONS:
Drug: Plecanatide

SUMMARY:
Multi-center, open-label, long-term safety study

DETAILED DESCRIPTION:
This is a phase 3, multicenter, open-label, long-term safety and tolerability study of 6 mg daily dose of plecanatide administered orally. Patients who are Study Completers or Eligible Screen Failures whose eligibility is confirmed at the end of their participation in the double-blind plecanatide studies SP304203-04 or SP304203-05 will be enrolled.

Beginning on Day 1, patients will take one (1) plecanatide 6.0 mg tablet in the clinic and thereafter every morning with approximately 240 mL (8 ounces) of liquid, with or without meals.

Safety and tolerability assessments and patients' self-assessment of disease severity will be performed according to the Schedule of Assessments.

Patients who discontinue early from the study will undergo an Early Withdrawal (EW) visit within 5 days after stopping study drug.

ELIGIBILITY:
Inclusion Criteria:

Patients with documented diagnosis of IBS-C who:

* Completed plecanatide study SP304203-04 or SP304203-05, were compliant with the previous study's requirements, and did not experience any Serious Adverse Event (SAE) deemed related to study drug during the course of the previous study, OR
* Failed screening in study SP304203-04 or SP304203-05 due to diary noncompliance (an exclusion in the core study) or due to an administrative reason and is allowed to enter this study by notification from Sponsor or delegate.

Key Exclusion Criteria:

* Patient is unwilling or unable to: participate in the study for the required duration, understand and sign the informed consent form (ICF) and undergo all protocol related tests and procedures throughout the study.
* Female patient of childbearing potential with a positive urine pregnancy test on Day 1.
* Male and female patients of childbearing potential who do not agree to continue to use the method of birth control used in the core double-blind plecanatide study for the duration of this clinical trial.
* Patient has experienced a significant negative change in health status during the course of participation in the core double-blind plecanatide study or after completion of the study.
* In the opinion of the Investigator or Medical Monitor, it is not in the patient's best interest to participate in the study. The reason(s) for the patient's exclusion must be specified.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2272 (Actual)
Dates: Start 2016-01; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bulawski, Study Director — Bausch Health
Locations (204):
- United States (204):
  - Synergy Research Site, Athens, Alabama
  - Synergy Research Site, Birmingham, Alabama
  - Synergy Research Site, Dothan, Alabama
  - Synergy Research Site, Foley, Alabama
  - Synergy Research Site, Guntersville, Alabama
  - Synergy Research Site, Huntsville, Alabama
  - Synergy Research Site, Saraland, Alabama
  - Synergy Research Site, Chandler, Arizona
  - Synergy Research Site, Phoenix, Arizona
  - Synergy Research Site, Surprise, Arizona
  - Synergy Research Site, Tucson, Arizona
  - Synergy Research Site, Conway, Arkansas
  - Synergy Research Site, Glendale, Arkansas
  - Synergy Research Site, Little Rock, Arkansas
  - Synergy Research Site, Artesia, California
  - Synergy Research Site, Canoga Park, California
  - Synergy Research Site, Carmichael, California
  - Synergy Research Site, Chula Vista, California
  - Synergy Research Site, Corona, California
  - Synergy Research Site, Costa Mesa, California
  - Synergy Research Site, El Cajon, California
  - Synergy Research Site, Encino, California
  - Synergy Research Site, Foothill Ranch, California
  - Synergy Research Site, Fountain Valley, California
  - Synergy Research Site, Garden Grove, California
  - Synergy Research Site, Huntington Beach, California
  - Synergy Research Site, La Mesa, California
  - Synergy Research Site, La Mirada, California
  - Synergy Research Site, Laguna Hills, California
  - Synergy Research Site, Lancaster, California
  - Synergy Research Site, Lomita, California
  - Synergy Research Site, Long Beach, California
  - Synergy Research Site, Los Angeles, California
  - Synergy Research Site, North Hollywood, California
  - Synergy Research Site, Northridge, California
  - Synergy Research Site, Orange, California
  - Synergy Research Site, Placentia, California
  - Synergy Research Site, Riverside, California
  - Synergy Research Site, San Bernardino, California
  - Synergy Research Site, San Diego, California
  - Synergy Research Site, San Marino, California
  - Synergy Research Site, Sherman Oaks, California
  - Synergy Research Site, Thousand Oaks, California
  - Synergy Research Site, Colorado Springs, Colorado
  - Synergy Research Site, Denver, Colorado
  - Synergy Research Site, Lafayette, Colorado
  - Synergy Research Site, Bristol, Connecticut
  - Synergy Research Site, Hamden, Connecticut
  - Synergy Research Site, Atlantis, Florida
  - Synergy Research Site, Boca Raton, Florida
  - Synergy Research Site, Boynton Beach, Florida
  - Synergy Research Site, Bradenton, Florida
  - Synergy Research Site, Brandon, Florida
  - Synergy Research Site, Brooksville, Florida
  - Synergy Research Site, Clearwater, Florida
  - Synergy Research Site, Cutler Bay, Florida
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Fort Lauderdale, Florida
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Homestead, Florida
  - Synergy Research Site, Inverness, Florida
  - Synergy Research Site, Jacksonville, Florida
  - Synergy Research Site, Lauderdale Lakes, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Miami Lakes, Florida
  - Synergy Research Site, Miami Springs, Florida
  - Synergy Research Site, Naples, Florida
  - Synergy Research Site, North Miami Beach, Florida
  - Synergy Research Site, Orange Park, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Ormond Beach, Florida
  - Synergy Research Site, Oviedo, Florida
  - Synergy Research Site, Pembroke Pines, Florida
  - Synergy Research Site, Pinellas Park, Florida
  - Synergy Research Site, Port Orange, Florida
  - Synergy Research Site, St. Petersburg, Florida
  - Synergy Research Site, Tamarac, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, Atlanta, Georgia
  - Synergy Research Site, Marietta, Georgia
  - Synergy Research Site, Snellville, Georgia
  - Synergy Research Site, Blackfoot, Idaho
  - Synergy Research Site, Boise, Idaho
  - Synergy Research Site, Meridian, Idaho
  - Synergy Research Site, Blue Island, Illinois
  - Synergy Research Site, Chicago, Illinois
  - Synergy Research Site, Evanston, Illinois
  - Synergy Research Site, Evergreen Park, Illinois
  - Synergy Research Site, Hoffman Estates, Illinois
  - Synergy Research Site, Morton, Illinois
  - Synergy Research Site, Oak Lawn, Illinois
  - Synergy Research Site, Schaumburg, Illinois
  - Synergy Research Site, Brownsburg, Indiana
  - Synergy Research Site, Indianapolis, Indiana
  - Synergy Research Site, Topeka, Kansas
  - Synergy Research Site, Wichita, Kansas
  - Synergy Research Site, Madisonville, Kentucky
  - Synergy Research Site, Owensboro, Kentucky
  - Synergy Research Site, Baton Rouge, Louisiana
  - Synergy Research Site, Crowley, Louisiana
  - Synergy Research Site, Mandeville, Louisiana
  - Synergy Research Site, Marrero, Louisiana
  - Synergy Research Site, Metairie, Louisiana
  - Synergy Research Site, New Orleans, Louisiana
  - Synergy Research Site, Shreveport, Louisiana
  - Synergy Research Site, Annapolis, Maryland
  - Synergy Research Site, Baltimore, Maryland
  - Synergy Research Site, Hagerstown, Maryland
  - Synergy Research Site, Oxon Hill, Maryland
  - Synergy Research Site, Marlborough, Massachusetts
  - Synergy Research Site, Chesterfield, Michigan
  - Synergy Research Site, Flint, Michigan
  - Synergy Research Site, Wyoming, Michigan
  - Synergy Research Site, Jackson, Mississippi
  - Synergy Research Site, Port Gibson, Mississippi
  - Synergy Research Site, Chesterfield, Missouri
  - Synergy Research Site, Hazelwood, Missouri
  - Synergy Research Site, St Louis, Missouri
  - Synergy Research Site, Missoula, Montana
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Marlton, New Jersey
  - Synergy Research Site, Albuquerque, New Mexico
  - Synergy Research Site, Brooklyn, New York
  - Synergy Research Site, Great Neck, New York
  - Synergy Research Site, Hopewell Junction, New York
  - Synergy Research Site, Kew Gardens, New York
  - Synergy Research Site, New Windsor, New York
  - Synergy Research Site, New York, New York
  - Synergy Research Site, North Massapequa, New York
  - Synergy Research Site, Poughkeepsie, New York
  - Synergy Research Site, Asheboro, North Carolina
  - Synergy Research Site, Cary, North Carolina
  - Synergy Research Site., Charlotte, North Carolina
  - Synergy Research Site, Charlotte, North Carolina
  - Synergy Research Site, Davidson, North Carolina
  - Synergy Research Site, Fayetteville, North Carolina
  - Synergy Research Site, High Point, North Carolina
  - Synergy Research Site, Jacksonville, North Carolina
  - Synergy Research Site, Kinston, North Carolina
  - Synergy Research Site, Raleigh, North Carolina
  - Synergy Research Site, Salisbury, North Carolina
  - Synergy Research Site, Wilmington, North Carolina
  - Synergy Research Site, Winston-Salem, North Carolina
  - Synergy Research Site, Fargo, North Dakota
  - Synergy Research Site, Beavercreek, Ohio
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Columbus, Ohio
  - Synergy Research Site, Dayton, Ohio
  - Synergy Research Site, Englewood, Ohio
  - Synergy Research Site, Kettering, Ohio
  - Synergy Research Site, Mentor, Ohio
  - Synergy Research Site, Middleburg Heights, Ohio
  - Synergy Research Site, Oklahoma City, Oklahoma
  - Synergy Research Site, Portland, Oregon
  - Synergy Research Site, Lansdale, Pennsylvania
  - Synergy Research Site, Levittown, Pennsylvania
  - Synergy Research Site, Philadelphia, Pennsylvania
  - Synergy Research Site, Smithfield, Pennsylvania
  - Synergy Research Site, Anderson, South Carolina
  - Synergy Research Site, Gaffney, South Carolina
  - Synergy Research Site, Greer, South Carolina
  - Synergy Research Site, Rapid City, South Dakota
  - Synergy Research Site, Athens, Tennessee
  - Synergy Research Site, Chattanooga, Tennessee
  - Synergy Research Site, Fayetteville, Tennessee
  - Synergy Research Site, Franklin, Tennessee
  - Synergy Research Site, Hermitage, Tennessee
  - Synergy Research Site, Jackson, Tennessee
  - Synergy Research Site, Kingsport, Tennessee
  - Synergy Research Site, Knoxville, Tennessee
  - Synergy Research Site, Memphis, Tennessee
  - Synergy Research Site, Nashville, Tennessee
  - Synergy Research Site, Austin, Texas
  - Synergy Research Site, Beaumont, Texas
  - Synergy Research Site, Carrollton, Texas
  - Synergy Research Site, Channelview, Texas
  - Synergy Research Site, Dallas, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, Humble, Texas
  - Synergy Research Site, Lampasas, Texas
  - Synergy Research Site, McKinney, Texas
  - Synergy Research Site, Missouri City, Texas
  - Synergy Research Site, Plano, Texas
  - Synergy Research Site, Port Arthur, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Sugar Land, Texas
  - Synergy Research Site, Ogden, Utah
  - Synergy Research Site, Orem, Utah
  - Synergy Research Site, Sandy City, Utah
  - Synergy Research Site, St. George, Utah
  - Synergy Research Site, Charlottesville, Virginia
  - Synergy Research Site, Chesapeake, Virginia
  - Synergy Research Site, Fairfax, Virginia
  - Synergy Research Site, Lynchburg, Virginia
  - Synergy Research Site, Newport News, Virginia
  - Synergy Research Site, Norfolk, Virginia
  - Synergy Research Site, Richmond, Virginia
  - Synergy Research Site, Bellevue, Washington
  - Synergy Research Site, Spokane, Washington
  - Synergy Research Site, Charleston, West Virginia
  - Synergy Research Site, Kingwood, West Virginia
  - Synergy Research Site, Morgantown, West Virginia
  - Synergy Research Site, La Crosse, Wisconsin
  - Synergy Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Barish CF, Crozier RA, Griffin PH. Long-term treatment with plecanatide was safe and tolerable in patients with irritable bowel syndrome with constipation. Curr Med Res Opin. 2019 Jan;35(1):81-85. doi: 10.1080/03007995.2018.1527303. Epub 2018 Oct 9. PMID 30277094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects with IBS-C from SP304203-04 (NCT02387359), SP304203-05 (NCT02493452), and SP304-20212 (NCT01722318), and subjects that did not previously participate in any plecanatide study, were enrolled.
Groups:
- Plecanatide: Plecanatide 6.0 mg tablets
  Plecanatide
Period: Overall Study
Arm/Group | Plecanatide
Started | 2272
Completed | 1842
Not Completed | 430
Not completed — Adverse Event | 97
Not completed — Death | 1
Not completed — Lack of Efficacy | 39
Not completed — Lost to Follow-up | 101
Not completed — Non-compliance with study drug | 15
Not completed — Physician Decision | 6
Not completed — Pregnancy | 6
Not completed — Protocol Violation | 18
Not completed — Withdrawal by Subject | 136
Not completed — Non-compliance with visits | 6
Not completed — Site closure | 4
Not completed — Subject moved | 1

BASELINE CHARACTERISTICS:
Arm/Group | Plecanatide
Number analyzed (Participants) | 2272
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1744
  Male | 528
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 504
  White | 1692
  More than one race | 13
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meters squared] — Population: Participants with height and weight information are included.
  kilograms per meters squared
    number analyzed (Participants) | 2269
    (all) | 28.4 (4.87)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Number of participants with adverse events with evidence to suggest a causal relationship between treatment and study drug.
Time Frame: up to 53 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Plecanatide
Number analyzed (Participants) | 2272
Participants | 205

ADVERSE EVENTS:
Time Frame: Up to 53 weeks.
Arm/Group | Plecanatide
All-Cause Mortality (participants affected / at risk) | 1/2272
Serious Adverse Events (participants affected / at risk) | 45/2272
Other Adverse Events (participants affected / at risk) | 341/2272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide (N=2272)
Alanine Aminotransferase Increased (Investigations) | 6 (6)
Aspartate Aminotransferase Increased (Investigations) | 5 (5)
Liver Function Test Abnormal (Investigations) | 1 (1)
Transaminases Increased (Investigations) | 1 (1)
Diverticulitis (Infections and infestations) | 3 (3)
Bacterial Pyelonephritis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridial Infection (Infections and infestations) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1)
Subcutaneous Abscess (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 (2)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm Fracture (Injury, poisoning and procedural complications) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Unstable (Cardiac disorders) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plecanatide (N=2272)
Diarrhoea (Gastrointestinal disorders) | 153
Nausea (Gastrointestinal disorders) | 29
Upper Respiratory Tract Infection (Infections and infestations) | 43
Urinary Tract Infection (Infections and infestations) | 34
Nasopharyngitis (Infections and infestations) | 34
Sinusitis (Infections and infestations) | 23
Headache (Nervous system disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02706483/Prot_SAP_000.pdf